CLINICAL TRIAL: NCT06707831
Title: Investigation of the Feasibility of the Trunk and Upper Extremity Assessments Used in the Scope of the ICF for Tele-Assessment in Children with Hemiplegic Cerebral Palsy
Brief Title: Feasibility of the Trunk and Upper Extremity Assessments for Teleassessment in Children Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Sefa Üneş, Assistant Professor, Hacettepe University
Other Study IDs: teleassessmentforCP
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Cerebral Palsy (CP)
Keywords: teleassessment; telerehabilitation; trunk and upper extremity; cerebral palsy; reliability and validity
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Study sample: Children with hemiplegic cerebral palsy aged 4 to 18 years
  Interventions: Other: Teleassessment

INTERVENTIONS:
Other: Teleassessment — Children underwent assessments on two occasions: one in face-to-face within a clinical setting, and the other through teleassessment using video conferencing. This video conference session was recorded to be later reviewed and scored by two separate raters.

SUMMARY:
This study was conducted to investigate the suitability of trunk and upper extremity assessments used within the scope of the ICF for tele-assessment in children with hemiplegic cerebral palsy (CP).

DETAILED DESCRIPTION:
A total of 36 children aged between 4-18 years with hemiplegic CP and their parents were included in the study. Children underwent evaluations on two occasions: one in face-to-face within a clinical setting, and the other through tele-assessment using video conferencing. This video conference session was recorded to be later reviewed and scored by two separate evaluators. For the assessment, the Trunk Control Measurement Scale (TCMS) was used for trunk control, the Upper Limb Physician Rating Scale (ULPRS) for upper extremity joint movement, the Upper Limb Selective Control Scale (SCUES) for selective ability, and the Quality of Upper Extremity Skills Test (QUEST) for skill quality. The bilateral hand use of children was assessed using the Abilhand-Kids, hemiplegic hand use with the Pediatric Motor Activity Log (PMAL), participation levels using The Assessment of Life-Habits (Life-H), and environmental factors were assessed using the European Child Environment Questionnaire (ECEQ), both face-to-face and through online surveys sent to families. Intra- and inter-rater reliability was determined by Intraclass Correlation Coefficient (ICC) and internal consistency was determined by Cronbach alpha coefficient (a). To determine validity, known group validity was examined based on the functional levels of children and concurrent validity was examined based on face-to-face assessment results. It was found that the internal consistency and both the intra- and inter-rater reliability of the TCMS (ICC: 0.82-0.91, p<0.05; α: 0.88-0.91), SCUES (ICC: 0.93-0.97, p<0.05; α: 0.93-0.94), ULPRS (ICC: 0.90-0.96, p<0.05; α: 0.94-0.95), and QUEST (ICC: 0.86-0.93, p<0.05; α: 0.93-0.94), conducted through both face-to-face assessment and tele-assessment by a physiotherapist or under supervision of a physiotherapist, were high to excellent. It was found that the tele-assessment reliability of Abilhand-Kids (ICC: 0.707, p<0.05) and PMAL (ICC: 0.60-0.70, p<0.05) was moderate; whereas, Life-H (ICC: 0.24) and ECEQ (ICC: 0.311) were determined to be weak. As a result, it was found that TCMS, SCUES, ULPRS, QUEST, Abilhand-Kids, and PMAL are suitable, valid, and reliable methods for tele-assessment; whereas, ECEQ and Life-H are not suitable for tele-assessment. These findings might partially diminish the necessity for the evaluation of children with CP in clinical settings, opening the way for suitable assessment methods. By ensuring equal opportunities for children with CP who cannot physically reach the clinic due to various reasons, reliable assessments can be conducted, contributing to the development of personalized tele-rehabilitation programs for the child. Although more extensive studies will be needed in the future, we expect transport costs to fall.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral (hemiplegic) cerebral palsy
* Being 4 - 18 years old
* Classified as Communication Function Classification System (CFCS) level 1 or 2
* Classified as Visual Function Classification System (VFCS) level 1 or 2
* Parents are able to read and write in Turkish

Exclusion Criteria:

* Diagnosed with epilepsy and active seizures in addition to CP
* Unable to use video call methods
* Refused to participate in the study
* Unable to co-operate during assessments
* The one who refused to continue with the assessments
* Those who had health problems during the assessments and could not continue the assessments

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cerebral palsy who visit the Pediatric Rehabilitation Department at Hacettepe University, Faculty of Physical Therapy and Rehabilitation, for routine treatment or examination.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Trunk Control Measurement Scale (TCMS) | 5 minutes
  The TCMS is a clinical tool used to assess trunk control in children with cerebral palsy. It evaluates both static and dynamic aspects of trunk control through tasks divided into three subscales: static sitting balance, dynamic sitting balance and dynamic reaching. It has total 15 items and each item is scored on a scale of 0 to 3, where higher scores indicate better trunk control. The total score ranges from 0 to 58, with subscale scores providing insights into specific components of trunk function.
Upper Limb Physician Rating Scale (ULPRS) | 5 minutes
  The ULPRS is a clinical assessment tool used to evaluate upper limb function in individuals with conditions like cerebral palsy. It focuses on assessing movement quality, range of motion, and functional use of the upper extremities during specific tasks or movements. The scoring typically reflects the severity of impairment, with lower scores indicating greater functional limitations. It is commonly used to monitor progress and guide treatment planning. Typically, items are scored individually, and the total score represents the overall severity of impairment or functionality.
Selective Control of Upper Extremity Scale (SCUES) | 5 minutes
  The SCUES is a clinical assessment tool designed to measure selective motor control in the upper extremities, particularly in individuals with neurological conditions such as cerebral palsy. It evaluates the ability to perform isolated, precise movements in the shoulder, elbow, wrist, and fingers without using compensatory patterns. Each limb is scored on a scale from 0 to 3 for each joint, where 0 indicates no selective movement and 3 indicates completely selective movement. The total score for a limb ranges from 0 to 15, with higher scores reflecting greater selectivity.
Quality of Upper Extremity Skills Test (QUEST) | 5 minutes
  The QUEST is a standardized tool designed to assess upper extremity function in children with neuromotor impairments, particularly cerebral palsy. It evaluates four domains: dissociated movements, grasp, protective extension, and weight-bearing, with 36 items scored from 0 (cannot perform) to 2 (performs fully). The scores are summed for each domain, and a total percentage score is calculated, with higher scores reflecting better movement quality and function. The QUEST is useful for guiding therapy and tracking progress over time.

SECONDARY OUTCOMES:
Abilhand-Kids | 5 minutes
  The Abilhand-Kids is a parent-reported questionnaire designed to assess manual ability in children with upper limb impairments, particularly those with cerebral palsy or other developmental disabilities. It measures the child's ability to perform daily activities requiring the use of both hands in a variety of functional contexts. The questionnaire includes 21 items, each rated on a 3-point scale: 0 (impossible), 1 (difficult), 2 (easy). The raw scores are converted to a linear Rasch scale, providing a standardized measure of manual ability. There is no fixed total score; instead, the Rasch analysis generates an overall ability estimate expressed in logits, allowing for comparison across individuals and groups. Higher scores represent the success in daily activities requiring the use of both hands.
Pediatric Motor Activity Log (PMAL) | 5 minutes
  The PMAL is a parent-reported assessment tool designed to measure the frequency and quality of motor activities performed by children with upper limb impairments, such as cerebral palsy. It focuses on how often and how well the child uses their affected arm in daily activities. It consists of 30 items, each rated on two scales: frequency and quality (both from 1 to 5). "Frequency" reflects how often the child uses their affected arm during specific activities, while "quality" reflects the child's ability to perform the activity. Scores for each item are summed to create a total score for both frequency and quality, with separate scores for each. Higher scores indicate better motor function, meaning the child uses their affected arm more frequently and with higher quality in daily activities. The total score is the sum of the frequency and quality scores, and higher
The Assessment of Life-Habits (Life-H) | 5 minutes
  The Life-H is a tool designed to evaluate the impact of a disability on an individual's ability to participate in daily life activities, covering various domains of life such as mobility, communication, social participation, and self-care. It is used across different age groups, including children and adults, with a variety of conditions, particularly those with physical or neurological impairments. Each item is scored on a scale from 0 to 9, where 0 indicates no difficulty, and 9 indicates complete difficulty or inability to perform the activity. The raw scores for each domain can then be converted to a standardized score ranging from 0 to 10. Higher scores indicate greater difficulty or more significant limitations in life habits. A higher total score reflects more challenges in daily life participation, while a lower score indicates better function and fewer limitations.
European Child Environment Questionnaire (ECEQ) | 5 minutes
  The ECEQ is a tool used to assess the impact of environmental factors on the participation and daily activities of children, particularly those with disabilities. It evaluates various environmental domains, including the home, school, and community, to determine how these settings either support or limit a child's ability to engage in everyday tasks. The ECEQ helps to identify barriers and areas where environmental modifications or supports may be needed to enhance the child's quality of life and participation.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rosenbaum P, Paneth N, Leviton A, Goldstein M, Bax M, Damiano D, Dan B, Jacobsson B. A report: the definition and classification of cerebral palsy April 2006. Dev Med Child Neurol Suppl. 2007 Feb;109:8-14. PMID 17370477
- [Background] Delioglu K, Unes S, Tuncdemir M, Ozal C, Biyik KS, Uzumcugil A. Interrater reliability of face-to-face, tele- and video-based assessments with the modified Mallet classification in brachial plexus birth injuries. J Hand Surg Eur Vol. 2024 May;49(5):576-582. doi: 10.1177/17531934231196118. Epub 2023 Sep 8. PMID 37684022
- [Background] Gungor F, Ovacik U, Ertan Harputlu O, Yekdaneh AA, Kurt I, Erturk Uzunoglu G, Polat Ilguz B, Akuzum F, Akbaba YA. Tele-assessment of core performance and functional capacity: Reliability, validity, and feasibility in healthy individuals. J Telemed Telecare. 2024 Jul;30(6):1017-1025. doi: 10.1177/1357633X221117335. Epub 2022 Aug 2. PMID 35916001
- [Background] Cabrera-Martos I, Ortiz-Rubio A, Torres-Sanchez I, Lopez-Lopez L, Rodriguez-Torres J, Carmen Valenza M. Agreement Between Face-to-Face and Tele-assessment of Upper Limb Functioning in Patients with Parkinson Disease. PM R. 2019 Jun;11(6):590-596. doi: 10.1002/pmrj.12001. Epub 2019 Mar 6. PMID 30840363
- [Background] Tan JR, Coulson S, Keep M. Face-to-Face Versus Video Assessment of Facial Paralysis: Implications for Telemedicine. J Med Internet Res. 2019 Apr 12;21(4):e11109. doi: 10.2196/11109. PMID 30977734
- [Background] Richmond T, Peterson C, Cason J, Billings M, Terrell EA, Lee ACW, Towey M, Parmanto B, Saptono A, Cohn ER, Brennan D. American Telemedicine Association's Principles for Delivering Telerehabilitation Services. Int J Telerehabil. 2017 Nov 20;9(2):63-68. doi: 10.5195/ijt.2017.6232. eCollection 2017 Fall. PMID 29238450
- [Background] Biyik KS, Ozal C, Tuncdemir M, Unes S, Delioglu K, Gunel MK. The functional health status of children with cerebral palsy during the COVID-19 pandemic stay-at-home period: a parental perspective. Turk J Pediatr. 2021;63(2):223-236. doi: 10.24953/turkjped.2021.02.006. PMID 33929112
- [Background] Yang P, Liu P, Li D, Zhao D. Corona Virus Disease 2019, a growing threat to children? J Infect. 2020 Jun;80(6):671-693. doi: 10.1016/j.jinf.2020.02.024. Epub 2020 Mar 3. PMID 32142929
- [Background] Rosenbaum PL, Silva M, Camden C. Let's not go back to 'normal'! lessons from COVID-19 for professionals working in childhood disability. Disabil Rehabil. 2021 Apr;43(7):1022-1028. doi: 10.1080/09638288.2020.1862925. Epub 2020 Dec 23. PMID 33355010
- [Derived] Unes S, Tuncdemir M, Ozal C, Delioglu K, Seyhan Biyik K, Kerem Gunel M. Tele-assessment of trunk control in children with cerebral palsy: Intra- and inter-rater reliability, and validity of the trunk control measurement scale. J Telemed Telecare. 2025 Apr 30:1357633X251336009. doi: 10.1177/1357633X251336009. Online ahead of print. PMID 40302488